CLINICAL TRIAL: NCT02757833
Title: Central Glutathione Levels in Women With Late Life Depression: a Cross Sectional Pilot Feasibility Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: A larger study collecting the same outcomes is currently being conducted by the study team.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10012689
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Female, Late Life Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Late Life Depressed Arm (Other): Participants in the Late Life Depressed arm will have a confirmed diagnosis of late-life depression.
  Interventions: Other: A 3 Tesla MRI scanner (Siemens, Erlangen Germany), will be used to measure levels of GSH in the brain.
- Healthy Control Arm (Other): Participants in the Healthy Control Arm will have no history of mental illness.
  Interventions: Other: A 3 Tesla MRI scanner (Siemens, Erlangen Germany), will be used to measure levels of GSH in the brain.

INTERVENTIONS:
Other: A 3 Tesla MRI scanner (Siemens, Erlangen Germany), will be used to measure levels of GSH in the brain. — Using the MEGA-PRESS pulse sequence, high resolution T1-weighted sagittal anatomic images covering the brain using an inversion-prepared MP-RAGE pulse sequence to produce high grey/white matter contrast will be acquired. These will be used to localize the spectroscopy voxel in the vmPFC. Magnetic field homogeneity will be optimized in the voxel using an automated map shimming procedure. MEGA-PRESS spectra will be acquired to detect the glutathione cysteinyl ß-CH2 peak at 2.95 ppm with the editing pulse set at the j-coupled a-CH resonance at 4.95 ppm. A reference unsuppressed water spectrum will be acquired for absolute quantification. Metabolite spectra will be fitted in the time domain using a Levenberg-Marquardt least squares minimization routine. The contribution of each metabolite to the in-vivo spectrum can be scaled to the water signal intensity from within the voxel of interest to obtain an absolute measurement of metabolite concentration.

SUMMARY:
Female participants with an episode of late-life depression (LLD) and age-matched control participants with no history of mental disorder will attend a one hour Magnetic Resonance Imaging (MRI). A 3 Tesla MRI scanner will be used to measure levels of glutathione (GSH) in the brain via magnetic resonance spectroscopy (1H MRS).

DETAILED DESCRIPTION:
This is a pilot/feasibility, single-centre, open-label, cross-sectional study. Research participants will be women aged 60 to 85. This study seeks to recruit 26 female participants; 13 participants with a confirmed diagnosis of late-life depression and 13 control participants with no history of mental illness. This pilot study will be used to determine if a larger Randomized Controlled Trial is feasible.

The role of antioxidant capacity in Late Life Depression (LLD) has thus far been inadequately assessed, providing the investigators with a timely opportunity to spearhead such an investigation. The results of this pilot study, and subsequent large-scale studies, will allow the investigators to identify novel targets for therapeutic intervention in LLD.

ELIGIBILITY:
Inclusion Criteria:

Late-life depression population inclusion criteria

* Patients in the LLD study arm will be females 60-85 years of age with a general good bill of health
* Patients in the LLD study arm will be presenting with mild to moderate MDD. Diagnosis of MDD will be confirmed through a Structured Clinical Interview for DSM-5-TR (SCID) Axis I disorder.
* LLD patients will have a Hamilton Depression Rating Scale (17-item version) score between 8-22
* LLD patients if being treated with any antidepressant agent, will be at a minimum of 4 weeks at therapeutic dosage of medication.

Healthy control (HC) population inclusion criteria:

* HC participants will be females between 60-85 years of age and in good general health
* HC participants will have no history of depression.

Exclusion Criteria:

* A primary diagnosis of any other mental health disorder (including substance dependence, post traumatic stress disorder, obsessive compulsive disorder, bipolar disorder, neurocognitive disorders, personality disorder, etc.)
* High risk of suicide as elicited by clinical interview
* History of head trauma
* History of severe vascular disease or cerebrovascular infarcts
* Any history of neurological disease (including Parkinson's disease or seizures)
* An ongoing acute episode of systemic inflammatory disease (e.g. rheumatoid arthritis, ulcerative colitis, crohn's disease)
* Any contraindications to MRI
* Additionally for Healthy Control participants only, a diagnosis of any mental health disorder

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Number of potential participants approached per month. | 2 years.
  At 2 years the number of potential participants approached per month will be calculated. This information will be used to determine if a larger Randomized Controlled Trial is likely to succeed.
Number of potential participants screened. | 2 years.
  At 2 years the number of potential participants screened will be assessed. This information will be used to determine if a larger Randomized Controlled Trial is likely to succeed.
Proportion of screened participants who enroll. | 2 years
  At 2 years the number of potential participants screened who enroll will be calculated. This information will be used to assess if a larger Randomized Controlled Trial is likely to succeed.
Rate of participant retention | 2 years
  At 2 years the rate of participant retention will be calculated. This information will be used to assess if a larger Randomized Controlled Trial is likely to succeed.
Cost per participant | 2 years
  At 2 years the cost per participant will be calculated. This information will be used to assess if a larger Randomized Controlled Trial is likely to succeed.
Quality of data available for analysis. | 2 years
  At 2 years the quality of the data available for analysis will be assessed. This information will be used to determine if a larger Randomized Controlled Trial is likely to succeed.

SECONDARY OUTCOMES:
Central glutathione levels in the brain | week 0
  Participants will attend only one assessment. During this assessment central glutathione levels in the brain will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No